CLINICAL TRIAL: NCT04206137
Title: Effects of Bilateral Asymmetrical Limbs Proprioceptive Neuromuscular Facilitation on Multifidus Muscle in Chronic Low Back Pain (CLBP)
Brief Title: Effects of Bilateral Asymmetrical Limbs Proprioceptive Neuromuscular Facilitation on Multifidus Muscle in CLBP.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Karachi (Other)
Responsible Party: Principal Investigator, Aftab Ahmed Mirza Baig,DPT, MSAPT, Principal Investigator, University of Karachi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: University of Karachi
Record Dates: First submitted 2019-12-15; First posted 2019-12-20 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Low Back Pain
Keywords: Muscle pain; Low Back Disorder; Exercise; Physical Therapy; Surface Electromyography
MeSH Terms: conditions — Low Back Pain; Myalgia; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (PNF rhythmic initiation group ) (Experimental): PNF rhythmic initiation with bilateral asymmetrical upper and lower limb pattern will administered on both sides, there will be 10 repetition and 3 sets for each side, 20 second rest between two sets.
  Interventions: Other: Group A (PNF rhythmic initiation group )
- Group B (Swiss ball exercise group) (Active Comparator): Swiss ball exercises will be administered. There will be 10 repetitions, with 5 sets, taking 15 seconds rest between each set.
  Interventions: Other: Group B (Swiss ball exercises)

INTERVENTIONS:
Other: Group A (PNF rhythmic initiation group ) — Lifting of arms and push the head back through the pattern of flexion -abduction-external rotation and neck in extension to the left in opposition of therapist hand resistance will be asked to do. At the end range of motion extensor muscles of back will start to contract.Then, reversing of that movement pattern to extension-adduction-internal rotation and neck flexion to right against the therapist resisting hands will be asked. this will be repeated on both sides
  Arms: Group A (PNF rhythmic initiation group )
Other: Group B (Swiss ball exercises) — Supine position: A ball will be placed under patient neck, and will be asked to bend hip and knee up to 90°. 5 times, 10 seconds hold Supine position: With a ball below the pelvis, knees bent, the ball press will be done with pelvis. 5 times, for 10 seconds hold.
  Crawling position: With a ball below one knee while keeping toes away from contact with the floor, the patient will balance first to stabilize the posture and slowly raise the other lower limb. This exercise will be performed in turn for the two lower limbs 10 times, with 10 seconds hold.
  Prone position: the patient will place a ball in front of pelvis and will repeatedly raise and lowered the two lower limbs alternately. There will be 10 repetitions, with 5 sets, taking 15 seconds rest between each set.
  Arms: Group B (Swiss ball exercise group)

SUMMARY:
The low back pain is a leading cause to limit individual functional activities worldwide and 60%-80% of adults are probable to get low back pain at least once in life time. Whereas, the chronic low back pain prevalence is 10%.The current literature suggests that any exercise is beneficial for reducing chronic nonspecific low back pain. This limits evidence regarding superiority of specific exercise for low back pain treatment. Therefore, a randomized control trial will be conducted at department of physiotherapy to assess which treatment is more effective in chronic low back pain at department of physiotherapy, institute of physical medicine and rehabilitation, Dow University of Health Sciences after synopsis approval. Overall 150 participants with 18-40 years old having chronic low back pain will be eligible and they will be included through non-probability, purposive sampling technique. The written informed consent will be taken from all the participants. They will be divided through systematic random sampling method into two groups, 75 in each group. Group A (experimental group) will receive Bilateral, asymmetrical limbs PNF pattern exercises and group B (control group) will receive Swiss ball exercises. All participants will be assessed using assessment form. Pain and functional disability will be measured by subjective outcome tools, visual analogue scale with 0-10cm and Oswestry disability index , respectively. Range of movement of lumbar and multifidus muscle activity will be measured by objective outcome tool, modified-modified Schober's test and surface electromyography, respectively. The pre & post treatment outcomes will be collected and recorded. Treatment sessions will be given thrice a week for 5 weeks. A maximum drop-out rate of 20% is expected. The Mean ± SD will be calculated for quantitative variables and frequencies and percentages for qualitative variables. The recorded outcome variables before and after the five weeks of treatment will be compared and analysed. The p-value of 0.05 will be considered as level of significant.

DETAILED DESCRIPTION:
Globally, Low back pain (LBP) is the commonest musculoskeletal pain, for which participants consult general practitioners. It is defined as "pain and discomfort, localized below the costal margin and above the inferior gluteal fold, with or without referred leg pain". The LBP with specific causes are rare (<15%). Whereas, majority (>80%) of LBP cases are non-specific LBP (NSLBP). The traditional temporal categorization comprises as acute LBP (<6 weeks), sub-acute LBP (≤12 weeks) or chronic LBP (>12 weeks). It is based on the duration of the current episode. The LBP is experienced in 60% to 80% of adults at some point in lifetime. There is 15% annual worldwide incidence rate of LBP and 30% point prevalence. LBP is one of the five leading causes of YLDS that contributes 57•6 million. The estimation suggests 5% to 10% of LBP cases will develop chronic. This chronicity is responsible for high treatment expenses, sick leave, and different sufferings.

The evidence based guidelines for LBP diagnosis suggest to first rule out any underlying pathology (spinal infection, cancer and fracture of spine and cauda equina syndrome). The LBP without any specific pathology is labelled as NSLBP. The routine use of radiologic imaging is not warranted based on clinical guidelines until presence of specific pathology. The goal of LBP treatment includes pain relief, function improvement, reduced work leave of absence, and chronicity prevention. The analgesics (topic or oral), exercise, manual therapy, traction, transcutaneous electrical nerve stimulation (TENS), back supports, acupuncture, biofeedback, spinal injections, and lastly, surgery may include in treatment options.Among exercise interventions the proprioceptive neuromuscular facilitation (PNF) exercise approach is designed to stimulate proprioceptors in order to enhance neuromuscular mechanism responses. The extremity patterns of PNF have diagonal direction with combination of movements, and these patterns are performed in line with the topographic arrangement of the muscles being used. Therefore, these exercises are thought to be suitable for muscles training anatomical-plane or anatomical-direction training programs. Moreover, PNF often have been used to improve the range of movement (ROM) and endurance. Various techniques of PNF training are used like rhythmic initiation, rhythmic stabilization, reversal of agonists, and reversal of antagonists.

In the existing literature there is little direction with mixed evidence to physiotherapists that what intervention is more beneficial to apply for CLPB. According to author's knowledge, the base to rely on PNF techniques needs evidence related to PNF patterns specification, that which lower limb PNF pattern is more effective. A randomized clinical trial will be conducted to explore the effects of bilateral, asymmetrical lower limb PNF patterns in flexion and in extension on multifidus in CLBP to evaluate and stabilize evidence based physical therapy practice in Pakistan.

Objectives:

1. To explore the effects of limbs PNF pattern exercises and Swiss ball exercises on multifidus motor activity, lumbar ROM, pain and functional disability in CLBP.
2. To determine the frequencies and statistical association of age, gender, body mass index (BMI) and occupation among participants in CLBP.
3. To determine the statistical association among multifidus motor activity, lumbar ROM, pain and functional disability of participants with CLBP before and after the exercise treatment.
4. T determine the effects of bilateral, asymmetrical limbs PNF pattern exercises and Swiss ball exercises in participants with CLBP
5. To compare the effects of bilateral, asymmetrical limbs PNF pattern exercises and Swiss ball exercises in participants with CLBP

Hypothesis:

1. Null hypothesis: There is no difference between effects of bilateral asymmetrical limbs proprioceptive neuromuscular facilitation and Swiss ball exercises on multifidus muscle in chronic low back pain.
2. Alternate Hypothesis: The effects of bilateral asymmetrical limbs proprioceptive neuromuscular facilitations are more beneficial than Swiss ball exercises on multifidus muscle in chronic low back pain.

Methodology:

Research design: The research design will be randomize control trial (RCT), experimental study.

Sampling technique: Non probability purposive sampling technique will be used. Sample size: Initially, a sample size of 54 human subjects was calculated through open epi software with 95% Confidence Interval and 80% power of test with post-test VAS mean (2.1) and standard deviation (0.85), in experimental group and post-test VAS mean (1.5) and standard deviation (0.69) in control group. Due to small sample size, it is increased to 150 with drop rate of 20%. The 75 participants per group will be considered.

Place of the study:

Physiotherapy department, Institute of physical medicine and rehabilitation (IPM&R), Dow University of Health Sciences (DUHS), Chand Bibi road, Karachi, Pakistan.

Data collection procedure:

After taking consent, the objectives of study will be told to all participants.The participants will be randomly allocated into two groups. All the participants will be assessed with outcome measures before after 5 weeks of intervention.

Interventions protocol: (half hour session, thrice a week for 5 weeks). Group A (experimental group) will receive, PNF rhythmic initiation with bilateral asymmetrical upper and lower limb pattern,

* The participant in supine position (on the back) with left arm in extension-adduction-internal rotation with right hand gripping his left wrist with right arm in modified extension-abduction-internal rotation. Neck will be in flexion looking at left hand.
* Therapist distal hand (hand away from head of the participant) will grip wrist of participant's left hand and the proximal hand (hand near to head of the participant) will be on top of the participant's head with fingers pointing towards the left side of participant neck.
* Participant will be asked to lift left arms and push the head back through the pattern of flexion -abduction-external rotation and neck in extension to the left in opposition of therapist hand resistance. At the end range of motion extensor muscles of back will start to contract.
* Then, participant will be asked to reverse the movement pattern to extension-adduction-internal rotation and neck flexion to right against the therapist resisting hands.
* It will be repeated on other side of participant.
* Then for lower limbs, participant's left leg will be in extension-abduction-internal rotation and right leg in extension-adduction-external rotation.
* Therapist will grasp the lateral and dorsal surfaces of both feet with distal hand. Proximal arm will be placed underneath the participant's thighs to hold them together.
* Then participant will be asked to lift both feet up, bend legs up and away towards right shoulder against therapist resistance.
* The right leg will go into flexion-abduction-internal rotation, the left leg into flexion-adduction-external rotation. At the end of range, the motion continues as lower trunk flexion with rotation and side-bending to the right.
* After that, participant will asked to reverse the left leg into extension-abduction-internal rotation and right leg in extension-adduction-external rotation against resistance. At end of range, the motion will carry on as trunk extension and elongation to the left with left rotation and side trunk flexion.
* It will be repeated on other side of participant.
* 10 repetition and 3 sets for each side, 20 second rest between two sets.

Group B (control group) will receive Swiss ball exercises :

1. Supine position: A ball will be placed under participant neck, and will be asked to bend hip and knee up to 90°. 5 times, 10 seconds hold
2. Supine position: With a ball below the pelvis, knees bent, the ball press will be done with pelvis. 5 times, for 10 seconds hold.
3. Crawling position: With a ball below one knee while keeping toes away from contact with the floor, the participant will balance first to stabilize the posture and slowly raise the other lower limb. This exercise will be performed in turn for the two lower limbs 10 times, with 10 seconds hold.
4. Prone position: Participant will place a ball in front of pelvis and will repeatedly raise and lowered the two lower limbs alternately. There will be 10 repetitions, with 5 sets, taking 15 seconds rest between each set.

Data analysis:

The Statistical package for the social sciences 21 version will be used for data analyzing. The mean and standard deviation will be calculated for quantitative variables like age. The qualitative variables will be shown through calculated frequencies and percentages. The outcome results of the study (decrease pain intensity, improve functional disability, improve range of movement and improve multifidus activity) taken before and after the treatment will be compared and analysed. The p-value of 0.05 will be considered as level of significant.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Low back pain (pain for > 3 month)

Exclusion Criteria:

* Any history related to spinal surgery
* Previous administration of epidural injections.
* Low Back Pain due to specific pathology,
* Neurological deficits (like stroke)
* Clinical disorder contraindicated to exercise.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-01-17 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | Change from baseline pain intensity at 5 weeks.
  The visual analogue scale is used for measurement of pain intensity. It is a continuous scale. It comprises a horizontal or vertical 10 centimeters or 100 millimeters line. The participant is asked to indicate a point of pain intensity by placing a line perpendicular to the Visual analogue scale line. The scale is most commonly referred by "no pain" with score of 0 and "worst imaginable pain" with score of 100 on the scale. The higher scores shows higher pain intensity and lower scores shows lower pain intensity.
Modified Modified Schober's test. | Change from baseline lumbar range of movement at 5 weeks.
  It is used during physical examination to assess the lumbar range of movement. It is highly co-related with lumbar range of movement measured through radiograph.
Surface electromyography | Change from baseline multifidus muscle activity at 5 weeks
  It is a record of the electrical activity associated with muscular contraction. The electromyography is recorded and the peak amplitude [maximal voluntary isometric contraction] is selected manually and recorded.

SECONDARY OUTCOMES:
Oswestry Disability Index | Change from baseline functional disability at 5 weeks
  It is a standard questionnaire with questions regarding pain and the disabling effect on daily activities. Its score ranges from 0 to 100 (no disability to maximum disability). Cut off value score "9" shows sensitivity 62% and specificity 55%.

CONTACTS AND LOCATIONS:
Overall Officials: Aftab Ahmed Mirza Baig, MSAPT, Principal Investigator — University of Karachi
Locations (1):
- Aftab Ahmed Mirza Baig, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bardin LD, King P, Maher CG. Diagnostic triage for low back pain: a practical approach for primary care. Med J Aust. 2017 Apr 3;206(6):268-273. doi: 10.5694/mja16.00828. PMID 28359011
- [Background] Ganesan S, Acharya AS, Chauhan R, Acharya S. Prevalence and Risk Factors for Low Back Pain in 1,355 Young Adults: A Cross-Sectional Study. Asian Spine J. 2017 Aug;11(4):610-617. doi: 10.4184/asj.2017.11.4.610. Epub 2017 Aug 7. PMID 28874980
- [Background] Meucci RD, Fassa AG, Faria NM. Prevalence of chronic low back pain: systematic review. Rev Saude Publica. 2015;49:1. doi: 10.1590/S0034-8910.2015049005874. Epub 2015 Oct 20. PMID 26487293
- [Background] Baig AAM, Ahmed SI, Ali SS, Rahmani A, Siddiqui F. Role of posterior-anterior vertebral mobilization versus thermotherapy in non specific lower back pain. Pak J Med Sci. 2018 Mar-Apr;34(2):435-439. doi: 10.12669/pjms.342.12402. PMID 29805422
- [Background] Metzger RL. Evidence-based practice guidelines for the diagnosis and treatment of lumbar spinal conditions. Nurse Pract. 2016 Dec 16;41(12):30-37. doi: 10.1097/01.NPR.0000508169.67852.bb. PMID 27820593
- [Background] Minghelli B, Oliveira R, Nunes C. Non-specific low back pain in adolescents from the south of Portugal: prevalence and associated factors. J Orthop Sci. 2014 Nov;19(6):883-92. doi: 10.1007/s00776-014-0626-z. Epub 2014 Aug 22. PMID 25145999
- [Background] Oliveira CB, Maher CG, Pinto RZ, Traeger AC, Lin CC, Chenot JF, van Tulder M, Koes BW. Clinical practice guidelines for the management of non-specific low back pain in primary care: an updated overview. Eur Spine J. 2018 Nov;27(11):2791-2803. doi: 10.1007/s00586-018-5673-2. Epub 2018 Jul 3. PMID 29971708
- [Background] Wells C, Kolt GS, Marshall P, Bialocerkowski A. The definition and application of Pilates exercise to treat people with chronic low back pain: a Delphi survey of Australian physical therapists. Phys Ther. 2014 Jun;94(6):792-805. doi: 10.2522/ptj.20130030. Epub 2013 Oct 31. PMID 24179139
- [Background] Luomajoki HA, Bonet Beltran MB, Careddu S, Bauer CM. Effectiveness of movement control exercise on patients with non-specific low back pain and movement control impairment: A systematic review and meta-analysis. Musculoskelet Sci Pract. 2018 Aug;36:1-11. doi: 10.1016/j.msksp.2018.03.008. Epub 2018 Mar 28. PMID 29631119
- [Background] Areeudomwong P, Buttagat V. Proprioceptive neuromuscular facilitation training improves pain-related and balance outcomes in working-age patients with chronic low back pain: a randomized controlled trial. Braz J Phys Ther. 2019 Sep-Oct;23(5):428-436. doi: 10.1016/j.bjpt.2018.10.005. Epub 2018 Oct 17. PMID 30361077
- [Background] Lee CW, Hwangbo K, Lee IS. The effects of combination patterns of proprioceptive neuromuscular facilitation and ball exercise on pain and muscle activity of chronic low back pain patients. J Phys Ther Sci. 2014 Jan;26(1):93-6. doi: 10.1589/jpts.26.93. Epub 2014 Feb 6. PMID 24567683
- [Background] French SD, Cameron M, Walker BF, Reggars JW, Esterman AJ. Superficial heat or cold for low back pain. Cochrane Database Syst Rev. 2006 Jan 25;2006(1):CD004750. doi: 10.1002/14651858.CD004750.pub2. PMID 16437495
- [Background] Noormohammadpour P, Kordi M, Mansournia MA, Akbari-Fakhrabadi M, Kordi R. The Role of a Multi-Step Core Stability Exercise Program in the Treatment of Nurses with Chronic Low Back Pain: A Single-Blinded Randomized Controlled Trial. Asian Spine J. 2018 Jun;12(3):490-502. doi: 10.4184/asj.2018.12.3.490. Epub 2018 Jun 4. PMID 29879777
- [Background] Shah SG, Kage V. Effect of Seven Sessions of Posterior-to-Anterior Spinal Mobilisation versus Prone Press-ups in Non-Specific Low Back Pain - Randomized Clinical Trial. J Clin Diagn Res. 2016 Mar;10(3):YC10-3. doi: 10.7860/JCDR/2016/15898.7485. Epub 2016 Mar 1. PMID 27134987
- [Background] Chiarotto A, Maxwell LJ, Terwee CB, Wells GA, Tugwell P, Ostelo RW. Roland-Morris Disability Questionnaire and Oswestry Disability Index: Which Has Better Measurement Properties for Measuring Physical Functioning in Nonspecific Low Back Pain? Systematic Review and Meta-Analysis. Phys Ther. 2016 Oct;96(10):1620-1637. doi: 10.2522/ptj.20150420. Epub 2016 Apr 14. PMID 27081203
- [Background] Kumar T, Kumar S, Nezamuddin M, Sharma VP. Efficacy of core muscle strengthening exercise in chronic low back pain patients. J Back Musculoskelet Rehabil. 2015;28(4):699-707. doi: 10.3233/BMR-140572. PMID 25467999
- [Background] Jeong JK, Kim YI, Kim E, Kong HJ, Yoon KS, Jeon JH, Kang JH, Lee H, Kwon O, Jung SY, Han CH. Effectiveness and safety of acupotomy for treating back and/or leg pain in patients with lumbar disc herniation: A study protocol for a multicenter, randomized, controlled, clinical trial. Medicine (Baltimore). 2018 Aug;97(34):e11951. doi: 10.1097/MD.0000000000011951. PMID 30142818
- [Background] Nowotny AH, Calderon MG, de Souza PA, Aguiar AF, Leonard G, Alves BMO, Amorim CF, da Silva RA. Lumbar stabilisation exercises versus back endurance-resistance exercise training in athletes with chronic low back pain: protocol of a randomised controlled trial. BMJ Open Sport Exerc Med. 2018 Nov 22;4(1):e000452. doi: 10.1136/bmjsem-2018-000452. eCollection 2018. PMID 30555717
- [Background] Chung S, Lee J, Yoon J. Effects of stabilization exercise using a ball on mutifidus cross-sectional area in patients with chronic low back pain. J Sports Sci Med. 2013 Sep 1;12(3):533-41. eCollection 2013. PMID 24149162
- [Derived] Baig AAM, Ansari B. Bilateral Asymmetrical Limb Proprioceptive Neuromuscular Facilitation Effects on Pain, Multifidus Activity, Range of Motion, and Disability in Low Back Pain: A Randomized Controlled Trial. J Manipulative Physiol Ther. 2022 Oct;45(8):604-613. doi: 10.1016/j.jmpt.2023.04.005. Epub 2023 Jun 9. PMID 37294220
- See also: Malla, S., Chahal, A., Tiku, R.K, Kaul B. Effect of motor control exercise on Swiss ball and PNF technique on non-specific low back pain. Health Sci .2018; 7(4):114-24 — https://www.ijmrhs.com/medical-research/effect-of-motor-control-exercise-on-swiss-ball-and-pnf-technique-on-non-specific-low-back-pain.pdf
- See also: Mavromoustakos, S., Beneka, A., Malliou, V., Adamidis, A., Kellis, E., Kagiaoglou, A., et al. Effects of a 6-week Proprioceptive Neuromuscular Facilitation Intervention on pain and disability in individuals with chronic low back pain. J Phys Act N. — https://www.panr.com.cy/article/effects-of-a-6-week-proprioceptive-neuromuscular-facilitation-intervention-on-pain-and-disability-in-individuals-with-chronic-low-back-pain/
- See also: Adler, S. S., Beckers, D., Buck, M. PNF in practice: an illustrated guide. Springer Science & Business Media. . 2007; https://doi.org/10.1007/978-3-540-73904-3 — https://link.springer.com/book/10.1007%2F978-3-540-73904-3
- See also: Osama, M., Mustafa, M. The prevalence of chronic low back pain and relative disability among farmers of swat. Int J Res Sci. 2017; 5(1), 37-42. — http://www.ijrs.org/ojs/index.php/IJRS/article/view/71/20